CLINICAL TRIAL: NCT00577889
Title: A Phase II Trial of 17-N-Allylamino-17-Demethoxygeldanamycin (17-AAG) in Combination With Gemcitabine in Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Gemcitabine Hydrochloride and Tanespimycin in Treating Patients With Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00156; MC0542; CDR0000445454 (Registry Identifier: PDQ (Physician Data Query)); N01CM17104 (NIH); NCT01647022 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2013-09

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (combination chemotherapy) (Experimental): Patients receive 750 mg/m2 gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and 154 mg/m2 tanespimycin IV over 1 hour on day 9 of course one. Beginning with course two (and for all subsequent courses), all patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and tanespimycin IV over 1 hour on days 2 and 9.
  Interventions: Drug: gemcitabine hydrochloride; Drug: tanespimycin
- Arm II (combination chemotherapy) (Experimental): Patients receive 750 mg/m2 gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and 154 mg/m2 tanespimycin IV over 1 hour on days 2 and 9 of course one. Beginning with course two (and for all subsequent courses), all patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and tanespimycin IV over 1 hour on days 2 and 9.
  Interventions: Drug: gemcitabine hydrochloride; Drug: tanespimycin
- Arm III (combination chemotherapy) (Experimental): Patients receive 750 mg/m2 gemcitabine hydrochloride IV over 30 minutes on day 8 and 154 mg/m2 tanespimycin IV over 1 hour on days 1 and 9 of course one. Beginning with course two (and for all subsequent courses), all patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and tanespimycin IV over 1 hour on days 2 and 9.
  Interventions: Drug: gemcitabine hydrochloride; Drug: tanespimycin

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 750 mg/m2 Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: tanespimycin — 154 mg/m2 Given IV
  Other Names: 17-AAG; 17-N-Allylamino-17-Demethoxygeldanamycin

SUMMARY:
This randomized phase II trial is studying three different schedules of gemcitabine hydrochloride and tanespimycin to see how well they work in treating patients with stage IV pancreatic cancer. Drugs used in chemotherapy, such as gemcitabine hydrochloride and tanespimycin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the effect of gemcitabine hydrochloride and tanespimycin (17-AAG) on 6-month survival rate in patients with stage IV pancreatic adenocarcinoma.

SECONDARY OBJECTIVES:

I. To determine the overall survival of these patients. II. To determine the time to disease progression (TTP) in these patients. III. To determine the confirmed response rate and duration of response in these patients.

IV. To determine the time to treatment failure in these patients. V. To determine the adverse events in these patients.

TERTIARY OBJECTIVES:

I. To determine the effects of treatment on molecular targets, such as CDK4, akt, phospho-akt, Hsp90, Hsp70, and CHK1, and correlate these with clinical endpoints, including survival at 6 months, TTP, response rate, and overall survival.

II. To determine the effect of gemcitabine hydrochloride metabolizing enzyme genotype on toxicity, and clinical outcome.

OUTLINE: This is a multicenter study. Patients are stratified according to Eastern Cooperative Oncology Group (ECOG) performance status (0, 1, or 2). Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8 and tanespimycin IV over 1 hour on day 9 of course one.

ARM II: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and tanespimycin IV over 1 hour on days 2 and 9 of course one.

ARM III: Patients receive gemcitabine hydrochloride IV over 30 minutes on day 8 and tanespimycin IV over 1 hour on days 1 and 9 of course one. Beginning with course two (and for all subsequent courses), all patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and tanespimycin IV over 1 hour on days 2 and 9.

Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Blood samples are collected at baseline and periodically during treatment for pharmacogenetic studies. Tumor tissue samples that are available are also collected for laboratory studies. Samples are analyzed for number of circulating tumor cells, levels of intracellular targets (e.g., CDK4, akt, phospho-akt, Hsp90, Hsp70, and CHK1), single nucleotide DNA polymorphisms, and Vav1 expression. Samples are analyzed by reverse transcriptase-polymerase chain reaction, immunofluorescence, and immunohistochemistry.

After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Clinical stage IV disease
* No known brain metastases
* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute Neutrophil Count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin normal
* Aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN (5 times ULN if liver metastases are present)
* Creatinine normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Ejection fraction > 40% by echocardiogram

  * Patients who received prior anthracyclines must have a normal ejection fraction by echocardiogram
* Corrected QT interval (QTc) < 500 msec
* Pulse oximetry > 88% on room air at rest and after gentle exercise (according to Group Medicare Guidelines)
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to tanespimycin (17-AAG) or gemcitabine hydrochloride
* No known allergy to eggs
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No active ischemic heart disease within the past 12 months
* No history of uncontrolled dysrhythmias
* No congenital long QT syndrome
* No left bundle branch block
* No other significant cardiac disease, including any of the following:

  * New York Heart Association class III or IV heart failure
  * Myocardial infarction within the past year
  * Poorly controlled angina
  * Uncontrolled dysrhythmias
  * History of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No clinically significant interstitial lung disease
* No symptomatic pulmonary disease requiring medication, including any of the following:

  * Dyspnea
  * Dyspnea on exertion
  * Paroxysmal nocturnal dyspnea
  * Significant pulmonary disease requiring oxygen*, including chronic obstructive/restrictive pulmonary disease
* No pulmonary or cardiac symptoms ≥ grade 2
* No history of cardiac or pulmonary toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or vincristine)
* No prior chemotherapy for metastatic disease
* No prior radiotherapy to the chest
* No prior radiotherapy that potentially included the heart in the field (e.g.,mantle radiotherapy)
* More than 3 months since prior adjuvant chemotherapy or chemotherapy for locally advanced disease
* More than 3 weeks since prior radiotherapy
* No concurrent medications that prolong or may prolong QTc
* No concurrent antiarrhythmic drugs
* No concurrent prophylactic colony-stimulating factors
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McWilliams, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 21 patients were accrued from May 30, 2008 to September 2, 2010.
Pre-assignment Details: A total of 21 patients were accrued and randomized onto one of 3 parallel arms (Arm I: 9 patients; Arm II: 6 patients; Arm III: 6 patients). One patient from Arm I canceled and was not used in baseline analysis nor endpoint analysis.
Period: Overall Study
Arm/Group | Arm I (Combination Chemotherapy) | Arm II (Combination Chemotherapy) | Arm III (Combination Chemotherapy)
Started | 9 | 6 | 6
Completed | 8 | 6 | 6
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One patient in Arm I canceled prior to treatment and was not used in baseline summary.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Combination Chemotherapy) | Arm II (Combination Chemotherapy) | Arm III (Combination Chemotherapy) | Total
Number analyzed (Participants) | 8 | 6 | 6 | 20
Age, Continuous [Median (Full Range); unit: years] | 59 [51 to 77] | 71 [51 to 81] | 67 [55 to 75] | 61.5 [51 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 5 | 4 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Six Month Survival Rate
Description: A patient that is alive at 6 months is considered a treatment "success". Estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I (Combination Chemotherapy) | Arm II (Combination Chemotherapy) | Arm III (Combination Chemotherapy)
Number analyzed (Participants) | 8 | 6 | 6
percentage of patients | 25 [7.5 to 83] | 67 [38 to 100] | 33 [11 to 100]

2. Secondary Outcome: Overall Survival Time
Description: Overall Survival time is defined as the time from registration to death due to any cause. Estimated using the method of Kaplan-Meier.
Time Frame: Assessed up to 2 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Combination Chemotherapy) | Arm II (Combination Chemotherapy) | Arm III (Combination Chemotherapy)
Number analyzed (Participants) | 8 | 6 | 6
months | 4.8 [2.8 to 6.6] | 6.9 [2.4 to 10.7] | 4.3 [1.9 to 15.3]

3. Secondary Outcome: Time to Disease Progression
Description: The time to disease progression is defined as the time from registration to the time of confirmed disease progression using the Response Evaluation Criteria In Solid Tumors (RECIST). Estimated using the method of Kaplan-Meier.
  Complete Response (CR): Disappearance of all target lesions and normalization of tumor biomarkers (CA 19-9 or CEA).
  Partial Response (PR): At least a 30% decrease in the sum of largest dimension(LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Time from registration to documentation of disease progression, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Combination Chemotherapy) | Arm II (Combination Chemotherapy) | Arm III (Combination Chemotherapy)
Number analyzed (Participants) | 8 | 6 | 6
months | 2.2 [1.4 to 4] | 4.1 [1.4 to 7.9] | 2.3 [1.4 to 4.0]

4. Secondary Outcome: Confirmed Response Rate
Description: A confirmed response is defined as a complete response (CR) or partial response (PR) observed in two consecutive evaluations at least 4 weeks apart using the Response Evaluation Criteria In Solid Tumors (RECIST). Estimated using the method of Kaplan-Meier.
  Complete Response (CR): Disappearance of all target lesions and normalization of tumor biomarkers (CA 19-9 or CEA).
  Partial Response (PR): At least a 30% decrease in the sum of largest dimension(LD) of target lesions taking as reference the baseline sum LD.Evaluated using RECIST criteria.
Time Frame: 2 consecutive evaluations at least 4 weeks, up to 6 courses of treatment
Measure: Number; unit: participants
Arm/Group | Arm I (Combination Chemotherapy) | Arm II (Combination Chemotherapy) | Arm III (Combination Chemotherapy)
Number analyzed (Participants) | 8 | 6 | 6
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Combination Chemotherapy) | Arm II (Combination Chemotherapy) | Arm III (Combination Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 6/8 | 2/6 | 2/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Combination Chemotherapy) (N=8) | Arm II (Combination Chemotherapy) (N=6) | Arm III (Combination Chemotherapy) (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Combination Chemotherapy) (N=8) | Arm II (Combination Chemotherapy) (N=6) | Arm III (Combination Chemotherapy) (N=6)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (22) | 4 (15) | 6 (16)
Abdominal pain (Gastrointestinal disorders) | 6 (13) | 5 (9) | 5 (10)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 1 (1) | 2 (2)
Gastric mucositis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (16) | 4 (8) | 5 (8)
Vomiting (Gastrointestinal disorders) | 4 (8) | 3 (4) | 3 (5)
Edema limbs (General disorders) | 1 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (24) | 5 (16) | 5 (15)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (6) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 4 (11) | 2 (9) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 4 (12) | 2 (3) | 3 (6)
Lymphocyte count decreased (Investigations) | 2 (6) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (7) | 4 (8) | 2 (5)
Platelet count decreased (Investigations) | 3 (7) | 2 (4) | 1 (1)
Weight loss (Investigations) | 1 (2) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 2 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (7) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less